CLINICAL TRIAL: NCT04342650
Title: Phase IIb Study to Evaluate the Efficacy and Safety of Chloroquine Diphosphate in the Treatment of Patients With Comorbidities, Without Severe Acute Respiratory Syndrome, Under the New Coronavirus (SARS-CoV2): a Double-blind, Randomized, Placebo-controlled Clinical Trial
Brief Title: Chloroquine Diphosphate in the Prevention of SARS in Covid-19 Infection
Acronym: CloroCOVID19II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundação de Medicina Tropical Dr. Heitor Vieira Dourado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE: 30504220.5.0000.0005
Record Dates: First submitted 2020-04-04; First posted 2020-04-13 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2020-07

CONDITIONS: COVID-19; SARS-CoV Infection; Severe Acute Respiratory Syndrome (SARS) Pneumonia; Clinical Trial
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Pneumonia | interventions — chloroquine diphosphate; Chloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): CQ 450mg twice daily (3 tablets of 150mg, every 12 hours) on day 1, followed by CQ 450mg once daily (3 tablets of 150mg) from D2 to D5. Oral administration.
  Interventions: Drug: Chloroquine Diphosphate
- Placebo (Placebo Comparator): Placebo tables of equal characteristics and duration of treatment.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Chloroquine Diphosphate — 150mg tablets Note: Tablets used in the study were Chloroquine Diphosphate (produced by Farmanguinhos/Fiocruz), and the dosing stated in the clinicaltrials.gov refers to chloroquine base (in mg).
  Other Names: chloroquine
  Arms: Intervention
Drug: Placebo oral tablet — 150mg placebo tablets
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled clinical trial. A total of 210 individuals aged over 18 years old, without a diagnosis of severe respiratory disease, who came to the study site with clinical and radiological suspicion of SARS-CoV2, will be randomized into two treatment groups at a 1:1 ratio to receive a 5-day CQ diphosphate tablets or placebo (tablet without active ingredient produced with the same physical characteristics).

ELIGIBILITY:
Inclusion Criteria:

1. Suspected cases of COVID-19, due to clinical and radiological data, during the epidemic;
2. Adult aged 18 or over, at the time of inclusion
3. Not having severe acute respiratory syndrome (SARS), that is, not using mechanical ventilation or supplemental oxygen, peripheral oxygen saturation> 94% in room air, and having a respiratory rate below 24 incursions per minute.
4. Patients with comorbidities only, due to the increased risk of developing SARS

Exclusion Criteria:

1. Patients with chronic use of drugs known to prolong QTc interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with onset of severe acute respiratory syndrome (SARS) | 7 days after randomization
  Evaluate if CQ diphosphate prevents the onset of SARS in patients on intervention group through standardized questionnaires.

SECONDARY OUTCOMES:
Mortality rate | after randomization, up to 28 days
  Mortality rate between intervention and placebo group on days 7, 14, and 28 after randomization
Number of participants in need of intensive care support | during and after intervention, up to 28 days
  Proportion of participants in need and duration of intensive care support after randomization
Viral concentration | After randomization, up to 7 days
  Viral load change in blood and oropharyngeal swab samples
Cumulative incidence of serious adverse events | During and after intervention, up to 28 days
  Incidence of serious adverse events during and after treatment
Cumulative incidence of grade 3 and 4 adverse events | During and after intervention, up to 28 days
  Incidence of grade 3 and 4 adverse events during and after treatment
Proportion of patients with discontinued treatment | after randomization, up to 28 days
  proportion of discontinuation or temporary suspension of treatment (for any reason)
Incidence of cardiac lesions | after randomization, up to 120 days
  proportion of patients with increased levels of troponin I
Incidence of cardiac disfunctions | after randomization, up to 120 days
  proportion and magnitude of QTcF interval increases higher than 500ms
Change in respiratory capacity | Day 120 after randomization
  Changes measured on day 120 will be compared to baseline, through spirometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital e Pronto Socorro Delphina Rinaldi Abdel Aziz, Manaus, Amazonas, Brazil

IPD SHARING:
Plan to Share IPD: Yes
all patient data will be shared after study publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: after study publication
Access Criteria: Upon formal request to researchers.